CLINICAL TRIAL: NCT01104571
Title: Effect of Perioperative AntiHER-2 Therapy on Early Breast Cancer Study - Biological Phase (EPHOS-B)
Brief Title: Trastuzumab or Lapatinib Ditosylate in Treating Women With Early Breast Cancer
Acronym: EPHOS-B
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: University of Manchester (Other); Manchester University NHS Foundation Trust (Other Government); Cancer Research UK (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000669882; ICR-CTSU-2008-10017 (Other: The Institute of Cancer Research Clinical Trials and Statistics Unit); UM-EPHOS-B; CRUK-08-002 (Other Grant/Funding Number: Cancer Research UK); MREC-09-H1208-52 (Other: Research Ethics Committee); ISRCTN-15004993 (Registry Identifier: ISRCTN); 2008-005466-30 (EudraCT Number); EU-21029
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Lapatinib; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1: Control (Other): No peri-operative therapy given
  Interventions: Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery
- Part 1: Trastuzumab (Experimental): Trastuzumab 6mg/kg iv given on days 1 & 8 pre-surgery & one dose of 2mg/kg iv between days 15-19 post surgery.
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy
- Part 1: lapatinib (Experimental): Lapatinib 1500mg/day p.o. continuously for 28 days. Should start 11 days (+2 or -1 day) before the scheduled surgery
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy
- Part 2: Control (Other): No peri-operative therapy
  Interventions: Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery
- Part 2: Trastuzumab (Experimental): Trastuzumab 6mg/kg iv given on days 1 & 8 pre-surgery & one dose of 2mg/kg iv between days 15-19 post surgery.
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy
- Part 2: lapatinib-trastuzumab combination (Experimental): Lapatinib 1000mg/day p.o. continuously for 28 days, in combination with trastuzumab 6mg/kg iv given on days 1 & 8 pre-surgery & one dose of 2mg/kg iv between days 15-19 post surgery. Both drugs should start 11 days (+2 or -1 day) before the scheduled surgery.
  Interventions: Biological: trastuzumab; Drug: lapatinib ditosylate; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: trastuzumab — Trastuzumab 6mg/kg iv given on days 1 & 8 pre-surgery & one dose of 2mg/kg iv between days 15-19 post surgery
  Arms: Part 1: Trastuzumab; Part 2: Trastuzumab; Part 2: lapatinib-trastuzumab combination
Drug: lapatinib ditosylate — Part 1: Lapatinib 1500mg/day p.o. continuously for 28 days. Should start 11 days (+2 or -1 day) before the scheduled surgery.
  Part 2: Lapatinib 1000mg/day p.o. continuously for 28 days. Should start 11 days (+2 or -1 day) before the scheduled surgery.
  Arms: Part 1: lapatinib; Part 2: lapatinib-trastuzumab combination
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
  Arms: Part 1: Trastuzumab; Part 1: lapatinib; Part 2: Trastuzumab; Part 2: lapatinib-trastuzumab combination
Procedure: neoadjuvant therapy
  Arms: Part 1: Trastuzumab; Part 1: lapatinib; Part 2: Trastuzumab; Part 2: lapatinib-trastuzumab combination
Procedure: therapeutic conventional surgery — therapeutic conventional surgery
  Arms: Part 1: Control; Part 2: Control

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether trastuzumab or lapatinib ditosylate is more effective in treating women with early breast cancer.

Update June 2013:

Since the initial development of EPHOS-B in 2007 more evidence in relation to safety and efficacy of anti-HER2 therapies are now available, and in particular, a growing body of evidence that combinations of two anti-HER2 therapies are more effective than monotherapies. Therefore this study has been amended (PART 2) to a 1:1:2 ratio to control, perioperative trastuzumab or the combination of lapatinib and trastuzumab.

PURPOSE: This randomized phase III trial is studying trastuzumab to see how well it works compared with lapatinib ditosylate (and in since June 2013 - compared with a combination of lapatinib and trastuzumab) in treating women with early breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether pre-operative treatment of HER-2 positive breast cancer patients with anti-HER2 therapy consisting of trastuzumab (Herceptin®) vs lapatinib ditosylate inhibits proliferation or increases apoptosis.
* To compare the effects of trastuzumab (Herceptin®), lapatinib ditosylate and the combination of lapatinib ditosylate and trastuzumab (Herceptin®) on the inhibition of proliferation or increase of apoptosis

Secondary

* To determine whether pre-operative anti-HER2 treatment reduces serum angiogenic factors.
* To identify molecular predictors of biological response to anti-HER2 therapy

OUTLINE:

This is a multicenter study.Patients are stratified according to center. Patients are randomized to 1 of 3 treatment arms.

PART 1: From Protocol versions 1 to 4:

* Arm I (control): Patients receive no neoadjuvant or adjuvant therapy. Approximately 14 days after randomization, patients undergo either breast-conservation surgery or mastectomy.
* Arm II (trastuzumab [Herceptin®]): Patients receive neoadjuvant trastuzumab IV over 90 minutes on days 1 and 8. Approximately 11 days after beginning of neoadjuvant therapy, patients undergo either breast-conservation surgery or mastectomy, and receive adjuvant trastuzumab on day 15.
* Arm III (lapatinib ditosylate): Patients receive neoadjuvant oral lapatinib ditosylate once daily on days 1-11. Within 24 hours after completion of neoadjuvant therapy, patients undergo either breast-conservation surgery or mastectomy, and receive adjuvant lapatinib ditosylate once daily on days 12-28.

Patients also receive standard adjuvant systemic therapy, including endocrine therapy (for hormone-sensitive disease) and/or chemotherapy and radiotherapy.

PART 2: From Protocol Version 5 (June 2013)

* Arm I (control): Patients receive no neoadjuvant or adjuvant therapy. Approximately 14 days after randomization, patients undergo either breast-conservation surgery or mastectomy.
* Arm II (trastuzumab [Herceptin®]): Patients receive neoadjuvant trastuzumab IV over 90 minutes on days 1 and 8. Approximately 11 days after beginning of neoadjuvant therapy, patients undergo either breast-conservation surgery or mastectomy, and receive adjuvant trastuzumab on day 15.
* Arm III (lapatinib ditosylate and (trastuzumab [Herceptin®] combination): Patients receive oral lapatinib ditosylate once daily on days 1-11. Within 24 hours after completion of neoadjuvant therapy, patients undergo either breast-conservation surgery or mastectomy, and receive adjuvant lapatinib ditosylate once daily on days 12-28. Patients also receive neoadjuvant trastuzumab IV over 90 minutes on days 1 and 8 and receive adjuvant trastuzumab on day 15.

PART 1 and 2:

Patients also receive standard adjuvant systemic therapy, including endocrine therapy (for hormone-sensitive disease) and/or chemotherapy and radiotherapy.

All patients undergo blood and tissue sample collection periodically for biomarker research studies comprising biomarkers of proliferation, apoptosis, and angiogenesis.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 10 years.

Peer Reviewed and Funded by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (by core biopsy) invasive breast cancer

  * Newly diagnosed disease
  * Resectable disease
* HER2-positive disease, defined as 3+ measured by IHC or gene amplification by fluorescent in situ hybridization (FISH)
* No evidence of metastatic disease (T4 category) or suspicion of distant metastases
* No inflammatory breast cancer
* Planned surgery within 1 month of diagnosis, and willing to undergo adjuvant chemotherapy and trastuzumab post-surgery
* Must consent to donation of tissue and blood samples
* Hormone receptor status known

  * Estrogen receptor-positive patients on hormone replacement therapy (HRT) must either continue HRT or must not have taken HRT within the past 3 weeks
  * Estrogen receptor-negative patients may enter the trial whether or not they have taken HRT within the past 3 weeks

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Serum creatinine < 2 times upper limit of normal (ULN) OR creatinine clearance > 30 mg/dL
* Bilirubin < 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* LVEF ≥ 55% by echocardiography or MUGA
* No clinically significant cardiac abnormalities or uncontrolled hypertension
* No prior myocardial infarction, heart failure, or significant angina
* No prior cancer at any other site that has been treated within the past 6 months (except basal cell carcinoma or cervical carcinoma in situ)
* No current active hepatic or biliary disease (except Gilbert syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease, per investigator assessment)
* No impaired gastrointestinal function that would sufficiently reduce lapatinib ditosylate absorption
* No known immediate or delayed hypersensitivity or reaction to drugs chemically related to trastuzumab or lapatinib ditosylate
* No altered mental state that would preclude obtaining written informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior trastuzumab (Herceptin®) therapy within the past 3 months
* No prior local cancer treatment (e.g., radiotherapy)
* No other concurrent investigational agent or anticancer therapy
* No use of herbal (alternative) therapies within 1 day of study entry (vitamin and/or mineral supplements allowed)
* No regular use of systemic steroids or other agents that could influence study endpoints (inhaled steroids allowed)
* No grapefruit and grapefruit juice for the duration of the study
* At least 14 days since prior and no concurrent CYP3A4 inducers
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 6 months since prior and no concurrent amiodarone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2010-04; Primary Completion 2017-08-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Increase in apoptosis, by change in the tumor (morphological apoptosis and activated caspase 3) measured at diagnosis and at surgery (biological phase) | 10-13 days
Fall in proliferation between diagnosis and surgery by change in proliferation measured by Ki67 immunohistochemical assessment (%) at diagnosis and at surgery (biological phase) | 10-13 days
Relapse-free survival (clinical phase) | TBC

SECONDARY OUTCOMES:
Changes in the angiogenic serum markers VEGF-A, VEGF R1, and CD105, measured at diagnosis, surgery (plus also tumor CD31) and 28-30 days post surgery (biological phase) | TBC
Pre-treatment and/or surgical expression of molecular markers (EGFR, Her-3, IGF1R, c-myc, AKT, p-ERK, pS6 inase, activated src, or truncated p95HER-2 expression) | TBC
Time to local recurrence (clinical phase) | TBC
Time to distant recurrence (clinical phase) | TBC
Overall survival (clinical phase) | TBC

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Bundred, Principal Investigator — Wythenshawe Hospital
Locations (1):
- Wythenshawe Hospital, Manchester, England, United Kingdom

REFERENCES:
- [Background] Bundred N, Cameron D, Armstrong A, Brunt AM, Cramer A, Dodwell D, Evans A, Hanby A, Hartup S, Hong A., Horgan K, Khattak I, Morden J, Naik J, Narayanan S, Ooi J, Shaaban A, Smith R, Webster-Smith M, Bliss J; on behalf of the EPHOS-B investigators. Effects of perioperative lapatinib and trastuzumab alone in combination in early HER2+ breast cancer - results from the EPHOS-B trial (CRUK/08/002). Eur J Cancer Supplements. 2016; 57 (Suppl 2): S5 #6LBA.
- [Background] Bliss JM, Robison LE, Webster-Smith MF, Emson MA, Kilburn LS, Smith IE, Robertson J, Dowsett M, Bundred NJ, Cameron DA, Vidya R, Horgan K, Evans AA, Kokan JS, Pinhel I, A'Hern R; on behalf of the POETIC and EPHOS-B Trialists. A trial model for the future in the search for personalised medicine - the UK POETIC and EPHOS-B perioperative trials experience. Cancer Res. 2011; 71(24 Suppl): Abstract number OT2-03-04.
- See also: Cancer Research UK - lay summary of EPHOS-B — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-effect-having-trastuzumab-or-lapatinib-before-surgery-early-breast-cancer-ephos-b
- See also: ISRCTN Registry — https://doi.org/10.1186/ISRCTN15004993